CLINICAL TRIAL: NCT02282358
Title: An Open-Label Phase II Study of Mocetinostat in Selected Patients With Mutations of Acetyltransferase Genes in Relapsed and Refractory Diffuse Large B-Cell Lymphoma and Follicular Lymphoma
Brief Title: Study of Mocetinostat in Selected Patients With Mutations of Acetyltransferase Genes in Relapsed and Refractory Diffuse Large B-Cell Lymphoma and Follicular Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: MethylGene Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-106
Record Dates: First submitted 2014-10-29; First posted 2014-11-04 (Estimated); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-05

CONDITIONS: Lymphoma; Relapsed and Refractory; Diffuse Large B-Cell Lymphoma and Follicular Lymphoma
Keywords: Mocetinostat; 14-106
MeSH Terms: conditions — Lymphoma; Recurrence; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — mocetinostat

ARMS (1):
- Mocetinostat (Experimental): Patients who harbor mutations for CREBBP and/or EP300 will be started on mocetinostat 70 mg orally three times per week on a 28 day schedule in cycle 1. The dose will be escalated in cycle 2 to 90 mg orally three times per week on a 28 day schedule if there are no grade 3 or higher drug related toxicities. Therapy will continue until disease progression, intolerable toxicities or death.
  Interventions: Drug: Mocetinostat

INTERVENTIONS:
Drug: Mocetinostat

SUMMARY:
The purpose of this study is to learn if the study drug mocetinostat can slow the progression of cancer in people who have a mutation in CREBBP or EP300 in the genetic makeup of their cancer. The potential side effects of mocetinostat will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patient has provided a signed study Informed Consent Form prior to performance of any study related procedurePatient is ≥ 18 years of age
* Patient has histologically confirmed diagnosis of diffuse large B cell lymphoma or follicular lymphoma harboring mutations in CREBBP or EP300 with relapsed or refractory disease
* Patients with diffuse large B cell lymphoma must have received at least two prior therapies and have received, declined or be ineligible for autologous or allogeneic stem cell transplant.
* Patients with follicular lymphoma must have received at least two prior therapies.
* Patients with either diffuse large B cell lymphoma or follicular lymphoma will be allowed to enroll after receiving only 1 prior therapy if they are felt to not be a candidate for further systemic chemotherapy.
* Patient has at least one measurable lesion (≥ 2 cm) according to Cheson criteria [45]. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 - Patient has adequate bone marrow and organ function by:

Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L

* Platelets ≥ 75 x 10^9/L (no platelet transfusion within past 14 days)
* Hemoglobin (Hgb) ≥ 9.0 g/dL (no RBC transfusion within past 14 days)
* International Normalized Ratio (INR) ≤ 1.5
* Serum Creatinine ≤ 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within 2.5 x ULN, or ≤ 5.0 x ULN for patients with documented hepatic involvement
* Serum bilirubin ≤ 1.5 x ULN or ≤ 3.0 x ULN for patients with Gilbert Syndrome or documented hepatic involvement.
* Patients must have fully recovered from major surgery and from the acute toxic effects of prior chemotherapy and radiotherapy (residual grade 1 toxicity, e.g. grade 1 peripheral neuropathy, and residual alopecia are allowed)

Exclusion Criteria:

* Patient has received previous treatment with HDAC inhibitors
* Patient has evidence of graft versus host disease (GVHD)
* Patient has active or history of central nervous system (CNS) disease
* Patient has impaired cardiac function including any of the following:
* Presence or history of pericardial effusion (definitions are provided in and/or pericarditis.
* Acute myocardial infarction, symptomatic angina pectoris ≤ 6 months prior to starting study drug
* Presence of congestive heart failure ≥ NYHA class 3
* QTc > 480 ms on a screening ECG
* Screening LVEF < 45% by echocardiography or MUGA
* Uncontrolled cardiac arrhythmia including uncontrolled atrial fibrillation/atrial flutter/sinus tachycardia, complete left bundle branch block, congenital long QT syndrome
* Presence of permanent cardiac pacemaker
* Other clinically significant heart disease
* Subject is taking warfarin at start of treatment or within 6 months prior to start of study treatment.
* Patient has a concurrent malignancy or has a malignancy within 3 years of study enrollment (with the exception of adequately treated basal or squamous cell carcinoma or nonmelanomatous skin cancer)
* Patient is concurrently using other approved or investigational antineoplastic agent
* Patient has received chemotherapy, targeted anticancer therapy, pelvic and/or para-aortic radiotherapy or has had major surgery ≤ 4 weeks (6 weeks for nitrosourea, monoclonal antibodies or mitomycin-C) prior to starting study drug or who have not recovered from side effects of such therapy
* Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of mocetinostat (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Patient is currently receiving increasing or chronic treatment (> 10 days) with corticosteroids or another immunosuppressive agent. The following uses of corticosteroids are permitted: single dose, topical applications (e.g., rash), inhaled sprays (e.g., obstructive airways diseases), eye drops or local injections (e.g., intra-articular).
* Patient has a history of non-compliance to medical regimen or inability to grant consent.
* Concomitant medications causing prolonged QT which cannot be discontinued or changed to a different medication prior to initiating study
* Patient is currently being treated with drugs known to be moderate or strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug. Patients must have discontinued strong inducers for at least one week and must have discontinued strong inhibitors before the start of treatment.

Note: the oral anti-diabetic drugs troglitazone and pioglitazone are CYP3A inducers.

* Patient has a known history of HIV (testing not mandatory), active Hepatitis B or C infection.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive serum hCG laboratory test (> 5 mIU/mL)
* Women of child bearing potential and men with reproductive potential, if they are unwilling to use adequate contraception while on study therapy and for 3 months thereafter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Zelenetz, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Mocetinostat: Participants who harbor mutations for CREBBP and/or EP300 will be started on mocetinostat.
Period: Overall Study
Arm/Group | Mocetinostat
Started | 7
Completed | 6
Not Completed | 1
Not completed — Nonevaluable | 1

BASELINE CHARACTERISTICS:
Arm/Group | Mocetinostat
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 67 [48 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Efficacy as Defined by Overall Response
Description: as defined by overall response rate of Mocetinostat at one year in patients with relapsed/refractory DLBCL and FL who have inactivating mutations of acetyltransferase genes. Response will be measured according to the 2007 revised Cheson criteria for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=50% decrease in sum of the product of the diameters (SPD) of up to 6 dominant lesions identified at baseline; Overall Response (OR) = CR + PR.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Mocetinostat
Number analyzed (Participants) | 7
Participants
  Partial Response | 1
  Stable Disease | 3
  Progression of Disease | 2
  Not Evaluable | 1

2. Secondary Outcome: Event Free Survival
Description: defined as time from the date of treatment start to the date of the first documented progressive disease (PD) or death due to any cause) rate using mocetinostat in this selected population will be estimated by the Kaplan-Meier method. Relapsed disease/progressive disease is defined as at least 50% increase of target measurable nodal lesions
Time Frame: up to 17.8 months
Measure: Median (Full Range); unit: months
Arm/Group | Mocetinostat
Number analyzed (Participants) | 7
months | 4.6 [0.3 to 17.8]

3. Secondary Outcome: Median Progression Free Survival/PFS
Description: is defined as the time from the date of first occurrence of CR or PR whichever is recorded first to the date of the first objectively documented progressive disease (PD) or death due to any cause. The duration of response will be assessed based on the sub-cohort of patients who showed responses also using Kaplan-Meier.
Time Frame: up to 17.8 months
Measure: Median (Full Range); unit: months
Arm/Group | Mocetinostat
Number analyzed (Participants) | 7
months | 4.6 [1.4 to 13.1]

4. Secondary Outcome: Number of Participants Evaluated for Toxicity According to the (NCI CTCAE) Version 4.0.
Description: will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Mocetinostat
Number analyzed (Participants) | 7
Participants | 7

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Mocetinostat 90 mg: Participants who harbor mutations for CREBBP and/or EP300 will be started on mocetinostat. The dose was escalated in cycle 2 to 90mg in the absence of DLTs.
Arm/Group | Mocetinostat 90 mg
All-Cause Mortality (participants affected / at risk) | 3/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mocetinostat 90 mg (N=7)
Enterocolitis Infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mocetinostat 90 mg (N=7)
Diarrhea (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Creatinine increased (Investigations) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Lethargy (Nervous system disorders) | 1
Lipase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Mucosal infection (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
White blood cell decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/58/NCT02282358/Prot_SAP_000.pdf